CLINICAL TRIAL: NCT05194085
Title: Kingasa Study: Interventions for Improved Post-partum ART Continuation and HIV Testing of Male Partners of Women in PMTCT B+ in Uganda
Brief Title: Impact of Male Provider Phone Calls to Increase Men's Clinic Linkage After HIVST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Monisha Sharma, Assistant Professor, School of Medicine: Global Health, University of Washington
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY0009286-A; 1K01MH115789-01A1 (NIH)
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: HIV; Linkage to Care; PMTCT; PrEP; ART Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Female SOC/Male SOC arm (No Intervention): Women will be provided the standard of care invitation letter for male partners for fast-track visit for HIV testing and laboratory HIV testing at enrollment and every 6 months until 6 months postpartum
- Female intervention/Male SOC arm (Active Comparator): Women will be provided the standard of care invitation letter for male partners for fast-track visit for HIV testing and POC VL tests for women at enrollment, delivery, and 6 months post-partum
  Interventions: Diagnostic Test: POC viral load testing
- Female SOC/Male intervention arm (Active Comparator): Women will be provided an invitation letter for male partners for wellness visits and laboratory-based HIV VL testing for women at enrollment, delivery, and 6 months post-partum
  Interventions: Other: Wellness visit services for male partners
- Female intervention/male intervention arm (Active Comparator): Women will be provided an invitation letter for male partners for wellness visits and POC viral load testing for women at enrollment, delivery, and 6 months post-partum
  Interventions: Diagnostic Test: POC viral load testing; Other: Wellness visit services for male partners

INTERVENTIONS:
Diagnostic Test: POC viral load testing — POC viral load testing- women randomized to have POC VL at enrollment, delivery and 6 months post-partum, will have a finger prick to obtain whole blood for the Cepheid Xpert HIV-1 RNA cartridge on the Xpert IV machine with results in 90 minutes. Women who are randomized to POC VL who have VL >200 c/ml will receive additional adherence counseling, following the STREAM protocol, [26] to address the challenges that they are having with ART use. At the delivery visit, infants of women in the POC VL arm will also have viral load testing done.
  Arms: Female intervention/Male SOC arm; Female intervention/male intervention arm
Other: Wellness visit services for male partners — Wellness visits for men- additional prevention services for men randomized to the intervention arm, including dual syphilis and HIV testing, blood pressure, visual acuity screening, and COVID-19 screening as part of wellness
  Arms: Female SOC/Male intervention arm; Female intervention/male intervention arm

SUMMARY:
Evaluate the impact of phone calls from a male counselor in increasing linkage to HIV care and PrEP among male partners of pregnant women attending PMTCT.

DETAILED DESCRIPTION:
Evaluate the impact of phone calls from a male counselor in increasing linkage to HIV care and PrEP among male partners of pregnant women attending PMTCT. Approach: Leveraging the staff and infrastructure of an ongoing study, Kingasa (R01MH113434), this study will evaluate the impact of phone calls from a male counselor to encourage male partners to link to HIV care or prevention services after HIV testing. The intervention will provide male counselor follow-up to 100 male partners of pregnant women in the intervention arm of the Kingasa study. Exit interviews will be conducted with men and their female partners to assess acceptability and challenges associated with the intervention. Outcomes assessed include ART initiation among HIV-positive men and PrEP by HIV-negative men at 6 months.

Hypothesis: The intervention of a phone call from a male counselor to provide counseling and encourage linkage to HIV care or prevention will be feasible and acceptable. It will result in a higher proportion of men linking to treatment and prevention compared to the standard of care arm of the Kingasa pilot study.

ELIGIBILITY:
Inclusion Criteria for women:

Age ≥18 or 14-17 years if an emancipated minor (pregnant or have a child), Currently pregnant, Not currently enrolled in an HIV treatment study, Male partner not known to be HIV-positive or has not tested in the past 3 months, Able and willing to provide written informed consent, Able and willing to provide adequate locator information for study retention purposes, Screening negative for any indication of intimate partner violence or social harm

Inclusion Criteria for men:

Female partner enrolled in Kingasa pilot study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Male partner linkage | 6 months from female partner enrollment
  To assess the proportion of HIV-negative male partners who initiate PrEP and HIV positive men who initiate ART among male partners who test for HIV and are provided male counselor phone follow up or who receive standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Monisha Sharma, PhD, ScM, Principal Investigator — University of Washington
Locations (1):
- Infectious Disease Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No